CLINICAL TRIAL: NCT06995521
Title: Use of Vorinostat as GVHD Prophylaxis in Children, Adolescents, and Young Adults With Non-Malignant Disorders Undergoing Allogeneic Blood and Marrow Transplantation
Brief Title: Vorinostat for Graft-versus-host Disease (GVHD) Prevention in Non-Malignant Adolescent and Young Adults (AYA) Population
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sung Won Choi (Other)
Responsible Party: Sponsor-Investigator, Sung Won Choi, Professor of Pediatrics, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00254327
Record Dates: First submitted 2025-05-12; First posted 2025-05-29 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-05

CONDITIONS: GVHD
Keywords: Non-malignant condition; Medication Vorinostat
MeSH Terms: interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vorinostat (Experimental): For matched sibling and matched unrelated donor transplant recipients Vorinostat will be given orally from day -10 to day 30 post-transplant.
  For Haploidentical donor transplant recipients Vorinostat will be given orally from day +5 (at least 24 hours after completion of the day +4 cyclophosphamide) through day 30 post-transplant.
  This will be given by liquid suspension or capsule by mouth.
  Interventions: Drug: Vorinostat

INTERVENTIONS:
Drug: Vorinostat — For Matched sibling and matched unrelated donor transplant recipients: Vorinostat will be given orally at a dose of 60 milligrams per square meter two times a day (BID) (120 mg/m2/day) from day -10 to day 30 post-transplant. The maximum dose will be 100 mg BID.
  Haploidentical donor transplant recipients:
  Vorinostat will be given orally at a dose of 60 mg/m2 BID (120 mg/m2/day) from day +5 (at least 24 hours after completion of the day +4 cyclophosphamide) through day 30 post-transplant. The maximum dose will be 100 mg BID.
  Dosing may be rounded by +/- 10%. Patients that are able to take capsules and whose calculated dose is ≥91 mg may take 100 mg capsules.
  Other Names: Zolinza

SUMMARY:
This is a single-arm, open label, phase 2 study to determine the safety and efficacy of vorinostat without serotherapy as GVHD prophylaxis when combined with either tacrolimus and methotrexate or post-transplant cyclophosphamide, tacrolimus, and mycophenolate in patients aged 1 to 26 years of age with non-malignant disorders undergoing bone marrow transplant following myeloablative conditioning.

DETAILED DESCRIPTION:
The Hypothesis of the trial:

The addition of vorinostat to standard GVHD prophylaxis without serotherapy will lead to improved GVHD-free event-free survival (GEFS) at 1-year post-transplant compared to historical serotherapy-containing GVHD prophylaxis regimens in patients with non-malignant disorders (NMD) undergoing Hematopoietic stem cell transplant (HSCT).

ELIGIBILITY:
Inclusion Criteria:

* Non-malignant condition amenable to transplantation, including but not limited to:

  1. Primary Immunodeficiency/Primary Immune regulatory disorders
  2. Inborn errors of metabolism
  3. Red blood cell disorders including hemoglobinopathies per protocol.
  4. Inherited bone marrow failure syndromes
* Available donor per protocol (matched siblings and matched unrelated donors, haploidentical donors). The use of mismatched unrelated donors will not be allowed for this study.
* Patient and/or legal guardian have signed the informed consent document
* Adequate organ function and performance status for allogeneic hematopoietic stem cell transplantation as defined by institutional practice:

  1. Pulmonary Function: diffusing capacity of the lungs for carbon monoxide (DLCO), forced expiratory volume in the first second (FEV1), Forced vital capacity (FVC) ≥50% predicted.
  2. Renal Function: Estimated or actual glomerular filtration rate (GFR) of ≥50 milliliters per minute (mL/min)/1.72 square meter (m2)
  3. Liver Function: aspartate aminotransferase (AST), alanine aminotransferase (ALT) <3x upper limit of normal; total bilirubin ≤2.5 milligrams per deciliter (mg/dL) unless related to disease or Gilbert syndrome. There is no upper limit for bilirubin in patients with confirmed Gilbert syndrome.
  4. Cardiac Function: Ejection fraction (EF) ≥50% or fractional shortening (FS) ≥26%
  5. Performance Status: Karnofsky/Lansky score ≥70%(HIV) and Human T-lymphotropic virus type (HTLV) I/II negative
  6. Infectious Disease testing: human immunodeficiency virus
* Patients with transfusion-dependent anemias (per protocol) should have a liver MRI to document hepatic iron content (certain values will be excluded)
* All patients of childbearing age must agree to practice 2 effective methods of contraception at the same time or agree to abstinence for 6 months after the last dose for females. Males with female sexual partners of reproductive potential should use contraception during treatment and for at least 3 months after the last dose.
* Patients treated with other investigational therapies for underlying disorder must discontinue these therapies prior to enrollment on the study unless, in the opinion of the treating physician, discontinuing these therapies prior to transplant would place the patient at undue risk of morbidity or mortality. In this case, patients must discontinue investigational therapies prior to initiation of the conditioning regimen.

Exclusion Criteria:

- Previous diagnosis of Fanconi anemia, dyskeratosis congenita or other telomere biology disorders, inherited genetic conditions known to adversely affect DNA-repair, or other disorders with known chemo- or radiosensitivity.

Additional testing may be conducted per investigator discretion but is not required for enrollment.

* Diagnosis of idiopathic severe aplastic anemia
* Diagnosis of severe combined immunodeficiency syndrome
* Diagnosis of malignancy within the last 5 years.
* Diagnosis of Epstein-Barr virus (EBV)-driven lymphoproliferative disorder within the last 5 years
* Uncontrolled bacterial, viral, or fungal infection at the time of enrollment
* Seropositive for HIV or HTLV
* Active hepatitis B or C
* Female patients that are pregnant or breast-feeding
* Inability to take oral medications.
* History of allergy to Vorinostat, related compounds, or any drugs used as part of the conditioning regimen or GVHD prophylaxis.
* Patients with transfusion-dependent anemia (≥8 packed red blood cell (PRBC) transfusions/year or ≥20 lifetime transfusions) that have a liver iron content of >8 milligram (mg) Iron(Fe)/Gram dry weight or evidence of bridging fibrosis or cirrhosis on biopsy.
* Patients enrolled on another GVHD-prevention clinical trial.
* Patients receiving an ex-vivo T cell-depleted or cluster of differentiation (CD34)-selected stem cell graft.
* Subjects that have had prior treatment with a histone deacetylase inhibitor (e.g. vorinostat, valproic acid) within the last 30 days.
* History of prolonged corrected QT interval (QTc) syndrome.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Ages: 1 Year to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
GVHD-free relapse-free Survival | 1 year
  Composite endpoint of 1-year GVHD-free, event free survival (GEFS) with the addition of vorinostat to standard serotherapy-free GVHD prophylaxis. Grade III-IV acute GVHD and chronic GVHD requiring immunosuppression will be considered in this assessment. Events contributing to this endpoint will include death due to any cause, primary or secondary graft failure/rejection, or second HSCT, whichever occurs first.
Primary graft failure/rejection | By day+42 post-Hematopoietic stem cell transplant
  Defined as never achieving an absolute neutrophil count (ANC) ≥500/microliters (µL) or never achieving ≥5% donor myeloid chimerism assessed by peripheral blood chimerism assays by day +42 post-Hematopoietic stem cell transplant (HSCT). Second infusion of hematopoietic stem cells is also considered indicative of primary graft failure by day +42 post-HSCT.
Secondary graft failure/rejection | Beyond day +42 post-HSCT
  Defined as <5% donor myeloid chimerism in peripheral blood beyond day +42 post-HSCT in patients with prior documentation of hematopoietic recovery with ≥5% donor cells by day +42 post-HSCT.
Secondary graft failure/rejection | By day +42 post-HSCT
  Second infusion of hematopoietic stem cells is also considered indicative of primary graft failure by day +42 post-HSCT

SECONDARY OUTCOMES:
Overall survival (OS) at day 100, 6-months, and 1-year post-HSCT | Day 100, 6-months, and 1-year post-HSCT
  This will be measured after HSCT.
Event Free Survival (EFS) at 1-year post-HSCT | 1 year post-HSCT
  An event will be defined as death due to any cause, graft rejection/failure, or second transplant, whichever occurs first.
Neutrophil engraftment at day 42 | Day 42 post-HSCT
  The time to engraftment of neutrophils >500/microliter (μl) was defined as per Center for International Blood and Marrow Transplant Research (CIBMTR) standards, requiring donor chimerism for neutrophil engraftment.
Platelet engraftment at day 100 post-HSCT | Day 100 post-HSCT
  Platelet engraftment is defined as independence from platelet transfusion for at least 3 days with a platelet count of more than ≥20 × 10^9/L.
Donor chimerism at day 28, 100, and 1-year post-HSCT | Day 28, 100, and 1-year post-HSCT
  Number of participants with full (95-100%), mixed (5-94%), and no (0-4%) donor cells. Chimerism is reported for unsorted whole blood and T cells.
Primary graft failure at day 42 | Day 42 post-HSCT
Secondary graft failure post-HSCT | Day 42 post-HSCT
Day 100 grade II-IV and grade III-IV GVHD | Day 100 post-HSCT
Chronic GVHD requiring immunosuppressive therapy (IST) at 1-year post-HSCT | 1-year post-HSCT
Incidence of grade 4 systemic infections (septicemia) at 1-year post-HSCT | 1-year post-HSCT
Incidence of viral reactivation by 1-year post-HSCT | 1 year post-HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Mark Vander Lugt, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No